CLINICAL TRIAL: NCT05595785
Title: The Effects of Yoga or Yoga Plus Mindfulness on Perceived Stress and Mindful Attention Awareness in a Chiropractic College Setting
Brief Title: Yoga Versus Yoga Plus Mindfulness on Perceived Stress and Mindful Attention Awareness in a Chiropractic College Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeanmarie R. Burke, PhD (Other)
Responsible Party: Sponsor-Investigator, Jeanmarie R. Burke, PhD, Dean of Faculty and Research, Northeast College of Health Sciences
Organization: Northeast College of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-01
Record Dates: First submitted 2022-10-15; First posted 2022-10-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Occupational Stress
Keywords: Yoga; Mindfulness; Stress; Psychological
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical-Based Yoga Practice (Experimental): Participants attended two 50-minute class sessions per week during the four week intervention phase.
  The physical-based yoga practice was Bishnu Ghosh lineage hatha yoga as taught by Mary Jarvis. The yoga class sessions included the physical postures of yoga with an emphasis on alignment, holding postures, and breathing normally.
  Each yoga class session sequentially included the following physical postures of yoga: (1) standing in stillness; (2) pranayama deep breathing and warm up; (3) standing series- balance postures, wide leg postures; (4) transition from the standing postures to the floor postures with tree pose; (5) floor series - wind removing, sit up movements, cobra posture, kneeling postures; (6) cool down-stretching, spine twist, Kapalbhati breathing, and Savasana.
  Interventions: Behavioral: Physical-Based Yoga Practice
- Mindfulness-Based Yoga Practice (Experimental): Participants attended two 50-minute class sessions per week during the four week intervention phase.
  The mindfulness-based yoga practice included all elements of the physical-based yoga class sessions with the addition of mindfulness cues.
  The mindfulness cues included body scan, mindful movement, and yoga nidra. Beyond verbal physical cues on how to control breathing and perform precise body movements during the yoga postures, verbal mindfulness cues asked participants to focus on the sensations of their breathing and body awareness non judgmentally, e.g. Feel your breathe move in through your nose and fill your lungs from bottom to top. Feel your breath exit the nose and empty lungs from top to bottom. Keep your attention on your breath and your body.
  Interventions: Behavioral: Mindfulness-Based Yoga Practice

INTERVENTIONS:
Behavioral: Physical-Based Yoga Practice — Physical-based yoga classes emphasized Bishnu Ghosh lineage hatha yoga. The 50 minute yoga classes were twice per week for four weeks. The yoga instructor had certifications in both Bikram and Amrit yoga practices and training in Bishnu Ghosh lineage hatha yoga as taught by Mary Jarvis
  Arms: Physical-Based Yoga Practice
Behavioral: Mindfulness-Based Yoga Practice — The mindfulness-based yoga classes included all elements of the physical-based yoga classes with the addition of mindfulness cues. The mindfulness cues included body scan, mindful movement, and yoga nidra. Certification of the instructor included the Integrative Amrit Method of Yoga Nidra that was inclusive of the use of mindfulness cues that coincided with the physical postures of yoga.
  Arms: Mindfulness-Based Yoga Practice

SUMMARY:
Objective: The purpose of the study was to compare the effects of different types of yoga practices on mindfulness and stress levels reported by students, faculty, and staff at a health professional school. Including mindfulness cues (body scan, mindful movement, and yoga nidra) with Bishnu Gosh lineage hatha yoga as taught by Mary Jarvis may have additive therapeutic effects on mindfulness and stress.

Methods: This was a quasi-experimental pre-post test design. Sixty-three individuals qualified for the study and were randomized in a 1:1 allocation ratio of matched pairs into either a physical-based yoga practice (Yoga Group, n = 31) or a mindfulness-based yoga practice (Yoga + Mindfulness Group, n = 32). Participants attended two 50-minute class sessions per week during the four-week intervention phase. The primary outcomes were the 10-item Perceived Stress Scale (PSS-10) and the 15-item Mindful Attention Awareness Scale (MAAS).

DETAILED DESCRIPTION:
Objective: The purpose of the study was to compare the effects of different types of yoga practices on mindfulness and stress levels reported by students, faculty, and staff at a health professional school. Including mindfulness cues (body scan, mindful movement, and yoga nidra) with Bishnu Gosh lineage hatha yoga as taught by Mary Jarvis may have additive therapeutic effects on mindfulness and stress.

Methods: This was a quasi-experimental pre-post test design. Sixty-three individuals qualified for the study and were randomized in a 1:1 allocation ratio of matched pairs into either a physical-based yoga practice (Yoga Group, n = 31) or a mindfulness-based yoga practice (Yoga + Mindfulness Group, n = 32). Participants attended two 50-minute class sessions per week during the four-week intervention phase. A sample size of 30 participants per class was deemed appropriate based upon the assumption of normality and the central limit theorem underlying the mathematics of inferential statistics.

The yoga class sessions included the physical postures of yoga with an emphasis on alignment, holding postures, and breathing normally. Throughout the yoga class session, the instructor demonstrated the performances of the physical postures. While participants were performing the physical postures, the instructor provided verbal alignment cues to the participants. As needed, the instructor also demonstrated postural modifications, which allowed all participants to perform all physical postures. Each class session sequentially included the following physical postures of yoga: (1) standing in stillness; (2) pranayama deep breathing and warm up; (3) standing series- balance postures, wide leg postures; (4) transition from the standing postures to the floor postures with tree pose; (5) floor series - wind removing, sit up movements, cobra posture, kneeling postures; (6) cool down-stretching, spine twist, Kapalbhati breathing, and Savasana.

The Yoga + Mindfulness class sessions included all elements of the yoga class session described above with the addition of mindfulness cues. The mindfulness cues included body scan, mindful movement, and yoga nidra. Beyond verbal physical cues on how to control breathing and perform precise body movements during the yoga postures, verbal mindfulness cues asked participants to focus on the sensations of their breathing and body awareness non judgmentally, e.g. Feel your breathe move in through your nose and fill your lungs from bottom to top. Feel your breath exit the nose and empty lungs from top to bottom. Keep your attention on your breath and your body. In general, the instructor reminded the participants throughout the Yoga + Mindfulness class session to "feel the sensation of ..."or "keep your attention on ..."as the instructor provided the alignment cues.

The primary outcomes were pre-post changes in the 10-item Perceived Stress Scale (PSS-10) and the 15-item Mindful Attention Awareness Scale (MAAS).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age Limits: from 20 years to 65 years of age

Exclusion Criteria:

* Pregnancy
* Nursing
* Wearing a pacemaker
* Prescription medications except for birth control or ADD/ADHD medications
* Stroke within the past three months
* Heart attack within the past three months
* Surgery within the past three months
* Car accident with injuries in the past three months
* Litigation of any type within the past three months or currently
* Currently participating in yoga activities once per week
* Currently participating in mindfulness activities once per week

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 1917-01-23 (Actual); Primary Completion 1918-01-22 (Actual); Study Completion 1918-01-22 (Actual)

PRIMARY OUTCOMES:
Changes in 10-Item Perceived Stress Scale | 4 weeks
  Perceived Stress Scale (PSS-10) is 10 item questionnaire that asks participants to rate their feelings and thoughts during the last month within the context of how often they felt or thought a certain way in different situations. The rating scale is 0 - never, 1 - almost never, 2 - sometimes 3 - fairly often 4 - very often. Classification system of stress levels included 0 to 13 as low stress, 14 to 26 as moderate stress and 27 to 40 as high stress.
Changes in 15-Item Mindful Attention Awareness Scale | 4 weeks
  The mindfulness domain was measured using the 15-item Mindful Attention Awareness Scale (MAAS). MAAS assesses an individual's dispositional mindfulness, which defines individual's awareness and attention during every day experiences, i.e. being present in the moment. The MAAS rates attention and awareness related to everyday experiences. MAAS numeric scale is 1- almost always, 2 - very frequently, 3 - somewhat frequently, 4, - somewhat infrequently, 5 - very infrequently, and 6 - almost never. The average numeric rating is the score on MAAS with higher mean values reflecting greater dispositional mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanmarie R Burke, PhD, Study Director — Northeast College of Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing includes study protocol, statistical analysis plan, and informed consent form upon e-mail request to Central Contact
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Until December 31, 2024
Access Criteria: e-mail Central Contact with request

REFERENCES:
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Taylor JM. Psychometric analysis of the Ten-Item Perceived Stress Scale. Psychol Assess. 2015 Mar;27(1):90-101. doi: 10.1037/a0038100. Epub 2014 Oct 27. PMID 25346996
- [Background] Cohen S, Janicki-Deverts D. Who's stressed? Distributions of psychological stress in the United States in probability samples from 1983, 2006, and 2009. J Appl Soc Psychol. 2012;42:1320-34.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Park T, Reilly-Spong M, Gross CR. Mindfulness: a systematic review of instruments to measure an emergent patient-reported outcome (PRO). Qual Life Res. 2013 Dec;22(10):2639-59. doi: 10.1007/s11136-013-0395-8. Epub 2013 Mar 29. PMID 23539467